CLINICAL TRIAL: NCT02845362
Title: Validation of the French Version of the Sydney Swallow Questionnaire in Patients With Neuromuscular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SSQVAL; 2016/18MAI/215 (Other: CEHF)
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Dysphagia; Neuromuscular Diseases
Keywords: Neuromuscular; dysphagia; Swallowing disorders; Questionnaire; Assessment
MeSH Terms: conditions — Deglutition Disorders; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dysphagia assessment (Experimental)
  Interventions: Other: Sydney Swallow Questionnaire

INTERVENTIONS:
Other: Sydney Swallow Questionnaire — The Sydney Swallow Questionnaire (SSQ) is a validated self-report symptom questionnaire, it contains 17 items recorded as visual analogue scales and is a tool specifically designed for evaluation of swallowing difficulties.

SUMMARY:
Measurements of dysphagia severity are important when making management decisions and in the objective evaluation of swallowing impairments. The Sydney Swallow Questionnaire (SSQ) is a validated self-report inventory using a visual analogue scale. This questionnaire permits a quantitative, sensitive, specific, repeatable and easily responsive evaluation of dysphagia in different pathology. Opposed to largely used videofluoroscopy swallowing study and endoscopy examinations, the SSQ is noninvasive, less expensive, avoids radiation exposure and enables a readily available assessment. Validated French version is not yet available. In the first phase of the study the investigators will validated this translation in dysphagic patients and control. Secondly, the investigators will validate the SSQ in Neuromuscular patients.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

Group 1:

* Healthy participants
* Able to speak, read and write in French
* Aged at least 18 years old

Group 2:

* Patients, with symptoms indicative of a deglutition disorder, referred for a videofluoroscopic study to the Otolaryngology, Head and Neck Surgery Department, Voice and Swallowing Clinic
* Able to speak, read and write in French
* Aged at least 18 years old

Phase 2:

* Clinical diagnosis of neuromuscular diseases
* Able to understand French

Exclusion Criteria:

Phase 1:

Group 1:

* History of neurological or neuromuscular disease
* History of any diagnosticated swallowing disorder

Group 2:

* Patients who could not be cataloged as dysphagic or non-dysphagic after the videofluoroscopic study evaluation
* Patients unable to answer the questionnaire

Phase 2:

* Patients who could not be cataloged as dysphagic or non-dysphagic
* Patients unable to answer the questionnaire

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Sydney Swallow Questionnaire | 10 minutes
  The participants were asked to fill out these questionnaires during the outpatient visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Audag, PT, Principal Investigator — Cliniques universitaires Saint-Luc, Brussels, Belgium
Locations (2):
- Belgium (2):
  - Cliniques universitaires Saint Luc, Brussels
  - Cliniques universitaires Saint-Luc, Brussels

IPD SHARING:
Plan to Share IPD: Undecided